CLINICAL TRIAL: NCT05300841
Title: The Effect of Pretreatment With Dydrogesterone Vs Combined Estradiol Valerate and Dydrogestrone on Clinical Pregnancy Outcome of ICSI in PCOS Patients"
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Ali, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSI in PCOS patients
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: PCOS; ICSI
MeSH Terms: interventions — Dydrogesterone; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dydrogesterone group (Active Comparator): Pretreatment with dydrogestrone (Duphaston, Abott Healthcare, Egypt) will be administered during the cycle preceding the ICSI cycle in a daily dose of 20 mg/ day starting 10 days before the presumed onset of menses
  Interventions: Drug: dydrogesterone 20 mg /d (Duphaston, Abott Healthcare , Egypt)
- Dydrogesterone plus estradiol valerate group (Active Comparator): will receive dydrogestrone 10mg /day plus estradiol valerate 2 mg /d (white tablets of cycloprognova, Bayer Schering, Germany) for 10 days.
  Interventions: Drug: dydrogesterone 20 mg /d (Duphaston, Abott Healthcare , Egypt); Drug: estradiol valerate 2 mg /d (white tablets of cycloprognova, Bayer Shering, Germany)

INTERVENTIONS:
Drug: dydrogesterone 20 mg /d (Duphaston, Abott Healthcare , Egypt) — Pretreatment with dydrogestrone (Duphaston, Abott Healthcare, Egypt) will be administered during the cycle preceding the ICSI cycle in a daily dose of 20 mg/ day starting 10 days before the presumed onset of menses
Drug: estradiol valerate 2 mg /d (white tablets of cycloprognova, Bayer Shering, Germany) — will receive dydrogestrone 10mg /day plus estradiol valerate 2 mg /d (white tablets of cycloprognova, Bayer Schering, Germany) for 10 days.
  Arms: Dydrogesterone plus estradiol valerate group

SUMMARY:
To analyze the effect of pretreatment with dydrogesterone vs combined estradiol valerate and dydrogesterone on embryologic parameters, chemical and clinical pregnancy rates of ICSI in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very common endocrine disorder affecting 5-7% of women in reproductive age. It is the leading cause of anovulatory infertility in this age group. It is characterized by ovulatory dysfunction, hyperandrogenism and polycystic ovary morphology on ultrasonography.

Assisted reproductive techniques (ART) are indicated when infertile women with PCOS are unable to become pregnant through standard ovulation induction methods. Many protocols have been used for ovulation induction in ICSI , GNRH agonist and GNRH antagonist protocols are the most commonly used nowadays. GNRH antagonist protocol use has been increased due to its high safety profile and progressive physician experience in controlled ovarian stimulation .

Steroid pretreatment is steroid administration in the cycle preceding the ICSI cycle. Due to oligo-menorrhea & unpredictability of menstruation in PCOS, steroid pretreatment is used to schedule the start of an ICSI cycle in women with PCOS. Also, it is expected to synchronize (homogenize) the follicular cohort, and thus increase both oocyte yield and gamete quality. Moreover, steroid pretreatment may have an impact on cycle outcome.

For these reasons, more attention has been paid to the potential interest of steroid pretreatments for scheduling GnRH antagonist cycles. Three main options have been used to achieve cycle programming. First the combined oral contraceptive pill (COCS)seems to be effective for scheduling menstruation but is not associated with increased oocyte yield . Furthermore, a meta-analysis pointed out that COCS pretreatment may be associated with fewer clinical pregnancies.Second, synthetic progestogens are good candidates because of their potent suppressive effect on pituitary gonadotrophin secretion and was associated with higher clinical pregnancy rate than COCS, placebo or no treatment. Finally, luteal administration of natural estrogens was proved to improve the synchronization of early antral follicle growth and to allow retrieval of two additional oocytes.

Either waiting for a spontaneous menses or using progestin is a better option than using COCs to induce menses in women with PCOS prior to ovarian stimulation using GnRH antagonist protocol for IVF. PCOS women using COCs had a lower live birth rate after fresh embryo transfer when compared with women using progestin for inducing menses or those with spontaneous menses. This difference, however, was not observed in the group who received an FET.

Dydrogesterone (DYD) is one of the synthetic forms of progesterone whose molecular structure and pharmacologic properties are closely related to endogenous progesterone .It is an orally active progestin that is non-thermogenetic, non-sedative and does not inhibit gonadotropin release and ovulation. It has weak antimineralocorticoid effects, negligible androgenic and glucocorticoid activities, and no antiandrogenic properties . Levonorgestrel (LNG) and Norgestrel (NG) are potent progestin exerting some androgenic activity, but no glucocorticoid or antimineralocorticoid properties .

Estradiol valerate is an estradiol ester, or a prodrug of estradiol. As such, it is an estrogen, or an agonist of the estrogen receptors. The affinity of estradiol valerate for the estrogen receptor is approximately 50 times lower than that of estradiol . In addition, estradiol valerate is rapidly cleaved into estradiol and is unable to reach target tissues in concentrations of significance, if at all .As such, estradiol valerate is essentially inactive in terms of estrogenic effect itself, acting solely as a prodrug to estradiol . Aside from dose adjustment to account for the difference in molecular weight, oral estradiol valerate is considered to be equivalent to oral estradiol. Because estradiol valerate is a prodrug of estradiol, it is considered to be a natural and bioidentical form of estrogen.

The current study aims to analyze the effect of pretreatment with dydrogestrone vs combined estradiol valerate and dydrogestrone on embryologic parameters, chemical and clinical pregnancy rates of ICSI for PCOS patients. The current study, being prospective and randomized, will differ from most of the previously conducted studies using steroid pretreatment in ICSI for PCOS patients. It also differs in comparing the pretreatment with dydrogesrone which is similar to natural progesterone with estradiol valerate which is similar to natural estradiol, together with Dydrogestrone.

ELIGIBILITY:
Inclusion Criteria:

* -Women with PCOS undergoing their first cycle of ICSI. PCOS diagnosis will be performed based on Rotterdam criteria (2003) based the presence of oligomenorrhea, polycystic ovaries on ultrasonography (defined as either an ovary that contains ≥ 12 antral follicles or ovarian volume>10cm3) as well as biochemical or clinical signs of hyperandrogenism, and after exclusion of other causes of hyperandrogenism as Cushing syndrome and CAH and hypothyroidism.
* age 18 to 35 years.
* BMI between 19 and 25 kg/square meter.
* AMH 3.5-6 ng/ml
* fresh or frozen embryo transfer

Exclusion Criteria:

* -FSH more than 12 IU /L
* AFC- performed on day 3 of the cycle- less than 4
* Existence of hydrosalpinx on ultrasonography
* uterine disorders as that caused by uterine fibroids.

  -. All male partners should have normal semen parameters .
* Women with more than 20 oocytes
* Any sign of early onset OHSS

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
chemical pregnancy rate | 6 gestational weeks
  positive pregnancy test in serum or urine without ultrasound evidence of a gestational sac; expressed per100 embryo transfer cycles.
Clinical pregnancy rate | 6 gestational weeks
  u/s visualization of a gestational sac and embryonic pole with heart beat expressed per per100 embryo transfer cycles.